CLINICAL TRIAL: NCT00916864
Title: Biomarker for Rapid Diagnosis of Hemispheric Stroke
Acronym: BE FAST!
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. Helmuth Steinmetz, Department of Neurology, Goethe-University, Frankfurt am Main, Germany
Other Study IDs: BEFAST!-1
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to estimate the diagnostic accuracy of a combined biomarker test (including NMDA-Receptor fragments [NR2-peptide] and Glial fibrillary acidic protein) used to differentiate between cerebral ischemia and intracerebral hemorrhage in patients with acute hemispheric stroke.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis
* at least one sign of cortical involvement (e.g., aphasia, neglect, gaze deviation, reduced level of consciousness)
* hospital admission within 4.5 hours after symptom onset

Exclusion Criteria:

* stroke/TIA within the last 3 months
* traumatic brain injury within the last 3 months
* history of brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with symptoms suspicious of acute hemispheric stroke to primary, secondary and tertiary care hospitals in Europe.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity and specificity for diagnosing cerebral ischemia and intracerebral hemorrhage) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Helmuth Steinmetz, MD, Study Chair — Department of Neurology, Goethe-University, Frankfurt, Germany
Locations (1):
- Department of Neurology, Goethe-University, Frankfurt am Main, Germany

REFERENCES:
- [Background] Dvorak F, Haberer I, Sitzer M, Foerch C. Characterisation of the diagnostic window of serum glial fibrillary acidic protein for the differentiation of intracerebral haemorrhage and ischaemic stroke. Cerebrovasc Dis. 2009;27(1):37-41. doi: 10.1159/000172632. Epub 2008 Nov 15. PMID 19018136
- [Background] Foerch C, Curdt I, Yan B, Dvorak F, Hermans M, Berkefeld J, Raabe A, Neumann-Haefelin T, Steinmetz H, Sitzer M. Serum glial fibrillary acidic protein as a biomarker for intracerebral haemorrhage in patients with acute stroke. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):181-4. doi: 10.1136/jnnp.2005.074823. Epub 2005 Sep 20. PMID 16174653
- [Background] Dambinova SA, Khounteev GA, Izykenova GA, Zavolokov IG, Ilyukhina AY, Skoromets AA. Blood test detecting autoantibodies to N-methyl-D-aspartate neuroreceptors for evaluation of patients with transient ischemic attack and stroke. Clin Chem. 2003 Oct;49(10):1752-62. doi: 10.1373/49.10.1752. PMID 14500616